CLINICAL TRIAL: NCT06549972
Title: Predictive Role of Early Blood KLK10 and Other Neuroinflammatory Molecules on Clinical Outcomes of Acute Ischemic Stroke
Brief Title: Predictive Role of KLK10 and Other Neuroinflammatory Molecules on Clinical Outcomes of AIS
Status: Completed | Type: Observational
Sponsor: Ruijin Hospital (Other)
Responsible Party: Principal Investigator, LI LONGXUAN, Professor, Ruijin Hospital
Other Study IDs: 2024092
Record Dates: First submitted 2024-08-06; First posted 2024-08-12 (Actual); Last update posted 2025-07-29 (Actual); Status verified 2025-07

CONDITIONS: Ischemic Stroke
MeSH Terms: conditions — Ischemic Stroke

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — For AIS patients, 10 ml of elbow venous blood will be collected at admission and then at 24 hours and 7 days after stroke onset. For healthy individuals, 10 ml of fasting elbow venous blood will be collected once. The dynamic changes and differential expression characteristics of a group of neuroinflammatory molecules, including KLK10, sTREM2, and GFAP in plasma will be observed.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- ischemic stroke group: The ischemic stroke group will be recruited from inpatients in the Department of Neurology at the Northern Campus of Ruijin hospital.
  Interventions: Other: Acute Ischemic Stroke
- control group (healthy individuals): The control group will be recruited from outpatient health check-up populations undergoing routine blood tests, biochemical tests, cranial CT, or MRI.

INTERVENTIONS:
Other: Acute Ischemic Stroke — first-ever anterior circulation AIS (Acute Ischemic Stroke)
  Groups: ischemic stroke group

SUMMARY:
This study aims to investigate the dynamic changes and differential expression characteristics of neuroinflammatory molecules such as kallikrein-related peptidase 10 (KLK10), soluble triggering receptor expressed on myeloid cells 2 (sTREM2), and glial fibrillary acidic protein (GFAP) in the plasma of patients with first-ever anterior circulation acute ischemic stroke (AIS). It will analyze the correlation between these molecules and the severity of neurological deficits, infarct volume, brain edema, hemorrhagic transformation, progressive stroke, and clinical outcomes at three months. The goal is to assess the predictive value of these molecules for AIS prognosis, guiding early treatment and new molecular targets for prevention and treatment.

DETAILED DESCRIPTION:
1. Informed Consent and Recruitment: Participants will be recruited based on inclusion and exclusion criteria.
2. divided two groups: the case group(ischemic stroke group) and the control group(healthy individuals).
3. First survey(At the time of admission): baseline Assessment- Survey on gender, age, medical history, smoking, drinking habits, and current medication; NIHSS score at admission; measurement of plasma levels of KLK10, sTREM2, and GFAP; a collection of blood glucose, creatinine, high-sensitivity C-reactive protein, blood cell analysis report, and brain MRI or CT imaging reports.
4. Second survey(24 hours after onset): NIHSS Score and Plasma Levels of KLK10, sTREM2, and GFAP Detection.
5. Third survey(Within 7 days of onset): Obtain brain CT or MRI reports to extract information on infarct volume, brain edema, and hemorrhagic transformation; perform NIHSS scoring to assess the occurrence of progressive stroke.
6. Forth survey( 3 months after onset): Final Assessment<if Good Functional Outcome or Mortality>:Record the Modified Rankin Scale (mRS) score at 3 months after stroke.

ELIGIBILITY:
Inclusion Criteria:

for AIS patients:

* Selection of 182 patients with first-ever acute ischemic stroke (AIS) who are hospitalized at our hospital, aged ≥18 years, with no restriction on gender;
* Patients must be admitted within 24 hours of the onset of AIS;
* Diagnosis must be confirmed by cranial magnetic resonance imaging (MRI) or computed tomography (CT);
* All enrolled patients must provide written informed consent.

for healthy controls:

* Age and gender-matched;
* No organic diseases;
* Written informed consent must be signed

Exclusion Criteria:

* Intracranial hemorrhage;
* Pregnancy;
* Stroke with unknown onset time;
* Malignant tumors;
* Hematologic disorders;
* Severe liver or kidney dysfunction;
* Recent myocardial infarction (less than 3 months);
* Ongoing anti-inflammatory drug treatment.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: A total of 182 patients with first-ever anterior circulation AIS (Acute Ischemic Stroke) hospitalized in the Neurology Department at the Northern Campus of our hospital will be selected as the observation group, and 91 healthy individuals undergoing physical examination will be chosen as the control group.
Sampling Method: Non-Probability Sample
Enrollment: 273 (Actual)
Dates: Start 2024-08-12 (Actual); Primary Completion 2025-06-30 (Actual); Study Completion 2025-06-30 (Actual)

PRIMARY OUTCOMES:
the Modified Rankin Scale (mRS) score | Record the Modified Rankin Scale (mRS) score at 3 months after stroke onset
  0 No symptoms.1 No significant disability; able to carry out all usual activities, despite some symptoms. 2 Slight disability; able to look after own affairs without assistance, but unable to carry out all previous activities. 3 Moderate disability; requires some help, but able to walk unassisted.4 Moderately severe disability; unable to attend to own bodily needs without assistance, and unable to walk unassisted. 5 Severe disability; requires constant nursing care and attention, bedridden, incontinent. 6 Dead.

SECONDARY OUTCOMES:
the mortality | Record mortality at 3 months after stroke onset
  mortality
the occurrence of hemorrhagic transformation | Record hemorrhagic transformation within 7 days after stroke onset
  based on brain CT scans to evaluate hemorrhagic transformation of cerebral infarction.
the occurrence of progressive stroke | Record progressive stroke within 7 days after stroke onset
  Neurological deficits are assessed using the NIHSS score. Progressive stroke is diagnosed if the NIHSS score increases by 2 points within 7 days after stroke onset.

CONTACTS AND LOCATIONS:
Overall Officials: Longxuan Li, Doctor, Principal Investigator — Ruijin Hospital Affiliated to Shanghai Jiao Tong University School
Locations (1):
- Neurology,Ruijin Hospital Affiliated to Shanghai Jiao Tong University School of Medicine, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2024-03-11): https://cdn.clinicaltrials.gov/large-docs/72/NCT06549972/Prot_SAP_000.pdf
  • Informed Consent Form (2024-03-11): https://cdn.clinicaltrials.gov/large-docs/72/NCT06549972/ICF_001.pdf